CLINICAL TRIAL: NCT06502184
Title: Functional and Mental Outcomes After Interdisciplinary Surgery for Patients With Obstructive Defecation Syndrome (ODS)
Brief Title: Mental Health Outcome After Surgery for Obstructed Defecation Syndrome (ODS)
Acronym: MentODSSurg
Status: Completed | Type: Observational
Sponsor: Evangelisches Klinikum Köln Weyertal gGmbH (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Claudia Rudroff, Head of the department of visceral surgery and functional surgery of the lower gastrointestinal tract, Evangelisches Klinikum Köln Weyertal gGmbH
Other Study IDs: Mental health in ODS Surgery
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Surgery; Obstructive Defecation Syndrome; Mental Health Issue; Depression/Anxiety; Outcomes
Keywords: mental health; depression; anxiety; obstructed defecation syndrome; surgery; bowel resection; rectopexy; outcome; follow up
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort of all patients who receive ODS surgery: laparoscopic resection rectopexy is performed

SUMMARY:
Background: Obstructed Defecation Synsdrome (ODS) causes people to strain and sometimes need help to go to the toilet. They think about going to the toilet a lot, which makes their lives worse. People with Obstructed Defecation Synsdrome (ODS) are more likely to be anxious and depressed than people with other illnesses.

Aim of the study: This study looked at how mental health affects Obstructed Defecation Synsdrome (ODS) patients before and after surgery.

DETAILED DESCRIPTION:
Aim, design, and setting of the study:

This study measures the mental burden of Obstructed Defecation Synsdrome (ODS) in patients scheduled for surgery for Obstructed Defecation Synsdrome (ODS) before and 6 months after surgery. The results are linked to how well the bowel works. All scores are checked before surgery and at 6 months after.

What do the investigators do to find this out ? The investigators look at patients' age, sex, body mass index (BMI), and other health problems. Defecation symptoms are measured using a validated questionnaire, the Altomare score, which has a maximum of 30 points. The rectal toxicity score reflects abdominal and bowel discomfort, which is determined by questions related to bowel dysfunction symptoms, such as diarrhea, meteorism, bleeding, and abdominal pain during bowel movement and defecation, and has a maximum of 32 points. The Wexner score is a 20-point questionnaire for fecal incontinence symptoms. Higher scores indicate greater severity of symptoms. Mental disorders are evaluated using the Personal Health Questionnaire 9 (PHQ-9) and General Anxiety Disorder 7 (GAD-7). Higher scores mean more severe symptoms.

Surgical procedure: For laparoscopic surgery under general anaesthesia, the patient is kept in a dorsal lithotomy position with their head down. The procedure opens the rectum, removes a part of the bowel and then rebuilds bowel continuity.

The investigators collect data on how long the operation took, how long the patient stays in hospital, and how many people have complications after the operation.

The scores will be reassessed at 6 months after surgery. For the clinical outcome, an improvement will be assumed at a reduction of 3 points and a strong improvement at a reduction of 6 points. Similarly, deterioration and major deterioration will be assumed at an increase of 3 points and 6 points. The results will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Obstructed Defecation Syndrome (ODS) scheduled for Surgery
* Conservative treatment failure
* Laparoscopic access possible

Exclusion Criteria:

• Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical and mental burdens of a consecutive group of patients, who is scheduled for surgery of Obstructed Defecation Syndrome (ODS) at the Evangelisches Klinikum Köln Weyertal, an academic teaching hospital associated with the university hospital cologne, which accommodates a tertiary pelvic organ and bowel dysfunction center as part of the surgical department, will be assessed before and 6 months after surgery.
  The self-reported clinical (bowel function) and mental score data are prospectively acquired as part of the standard operating procedure for all patients with functional bowel motility disorders in the investigators' hospital. Informed consent for the planned procedure, data collection, and publication of the results was obtained from all patients before surgery.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Mental Health Outcome - Depression | 6 months
  Depression in patients with Obstructed Defecation Syndrome (ODS) is measured with a questionnaire (score) before and after Surgery.
  The Personal Health Questionnaire 9 (PHQ-9) as an established score for depressive symptoms is used. It has a maximum of 27 points and higher scores mean a worse outcome. The score is divided into five subgroups of depression severity, namely, nonminimal (0-4 points), mild (5-9 points), moderate (10-14 points), moderately severe (15-19 points), and severe (20-27 points).
Mental Health Outcome - Anxiety | 6 months
  Anxiety in patients with Obstructed Defecation Syndrome (ODS) is measured with a questionnaire (score) before and after Surgery, as well, since this is another important outcome measure for mental health.
  Anxiety symptoms are measured by the General Anxiety Disorder 7 questionnaire (GAD-7), which has a maximum of 21 Points. Higher scores represent a higher burden and a worse outcome. GAD-7 is devided into four subgroups that differentiate the severity of anxiety into minimal (0-4 points), mild (5-9 points), moderate (10-14 points), and severe levels (15-21 points).

SECONDARY OUTCOMES:
Bowel Function - Altomare Score | 6 months
  Bowel function scores after Surgery for Obstructed Defecation Syndrome (ODS) before an after 6 months from surgery.
  Defecation symptoms were measured using the Altomare score, a validated ODS questionnaire with a maximum of 30 points. In the questionnaire higher scores indicate greater severity of symptoms. However, no validated cutoff levels exist for scoring.
Bowel Function - rectal toxicity score | 6 months
  Bowel function scores after Surgery for Obstructed Defecation Syndrome (ODS) before an after 6 months from surgery. The rectal toxicity score reflects abdominal and bowel discomfort, which is determined by questions related to bowel dysfunction symptoms, such as diarrhea, meteorism, bleeding, and abdominal pain during bowel movement and defecation, and has a maximum of 32 points. As for the Altomare score, for the rectal toxicity higher score values indicate greater severity of symptoms. However, no validated cutoff levels exist .
Bowel Function - Wexner incontinence score | 6 months
  The Wexner incontinence score is an established questionnaire for fecal incontinence symptoms, with a maximum of 20 points. It is measured before surgery and after 6 months follow up, as well. As for the other questionnaires, higher scores indicate greater severity of symptoms. However, no validated cutoff levels exist.

OTHER OUTCOMES:
Surgical Outcome | 6 months
  Morbiditiy and Mortality as measured by the Clavien Dindo Classification (CDC). The CDC distinguishes postoperative morbidity and mortality based on severity, which ranges from mild complications (CDC 1) and complications requiring medication (CDC 2) to complications requiring intervention in local anesthesia (CDC 3a) or narcosis (3b), septic complications (CDC 4a) combined with multiorgan failure (4b), and death (CDC 5). CDCs 1-3a are classified as minor complications, and CDCs 3b-4b are classified as major complications.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Rudroff, MD, Principal Investigator — Evangelisches Klinikum Köln Weyertal
Locations (1):
- Evanglisches Klinikum Koeln Weyertal, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Patients are not willing to share the data

REFERENCES:
- [Background] Rudroff C, Madukkakuzhy J, Hernandez AV, Otten J, Ulrici C, Karapanos L, Ludwig S. Early safety and efficiency outcomes of a novel interdisciplinary laparoscopic resection rectopexy combined with sacrocolpopexy for women with obstructive defecation syndrome and pelvic organ prolapse: a single center study. BMC Surg. 2024 Jun 14;24(1):185. doi: 10.1186/s12893-024-02474-4. PMID 38877450